CLINICAL TRIAL: NCT05632705
Title: A Randomised Trial to Evaluate the Efficacy and Feasibility of a Closing Pack to Reduce the Rate of Surgical Site Infection Following Caesarean Section
Brief Title: Efficacy of Using a Closing Pack to Reduce Postpartum Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, Leon Snyman, Prof, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PPS trial 2
Record Dates: First submitted 2021-03-08; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Prevention of Postpartum Sepsis

STUDY DESIGN:
Intervention Model Description: Randomised trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not have information with regards to the intervention arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): In this arm, prior to closing the sheath and skin, unused drapes, gloves and instruments will be used to close the sheath and the skin.
  Interventions: Other: Closing pack
- Control arm (No Intervention): In this arm sheath and skin closure will be according to the standard protocol

INTERVENTIONS:
Other: Closing pack — A closing pack, new sterile gloves and new sterile drapes will be used when commencing closure of the sheath and skin
  Arms: Intervention arm

SUMMARY:
Randomised trial comparing the efficacy and feasibility of using a sterile closing pack to reduce postpartum sepsis

DETAILED DESCRIPTION:
Pregnant patients meeting the inclusion criteria undergoing elective or emergency caesarean section will be eligible for recruitment. Patients will be randomised into two arms. In the control arm sheath and skin closure will be performed with the instruments used to perform the caesarean section, as per the current standard of care. In the intervention arm, after suturing the uterine incision and obtaining hemostasis and before commencing closure of the sheath and skin, the surgical team (obstetrician, assistant and scrub sister) will don clean sterile gloves, open clean sterile linen to drape on top of the existing linen and open a pack of clean sterile instruments to close the sheath and skin.

ELIGIBILITY:
Inclusion Criteria:

* women 18 years and older willing and able to provide consent

Exclusion Criteria:

* women who are not able or willing to provide consent patients with existing maternal infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients who are pregnant undergoing caesarean section
Enrollment: 1000 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy to reduce surgical site infections within seven days | Seven days post-operatively
  Incidence of surgical site infections in both arms

SECONDARY OUTCOMES:
Efficacy to reduce postpartum endometritis within seven days | Seven days post-operatively
  Incidence of postpartum endometritis in both arms
Feasibility of using a closure pack | At the time of caesarean section
  Assess the availability as well as use of the sterile closing pack

CONTACTS AND LOCATIONS:
Locations (1):
- Kalafong Provincial Tertiary Hospital, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No